CLINICAL TRIAL: NCT07067073
Title: ANTI-DYNAMIC LINE Test for Cream: A Mono-centric 8-week Clinical Evaluation on Facial and Neck Dynamic Wrinkles in Chinese Female Subjects Aged 18-35
Brief Title: ANTI-DYNAMIC LINE Test for Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C24005075
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dynamic Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Cream Arm (Experimental): Participants apply the investigational cream (Formula# 899675 44A) on the entire face and neck twice daily for 8 weeks following a 2-week wash-out period. Application is supervised on-site at baseline and self-administered at home thereafter. Clinical assessments and facial/neck image capture are conducted at baseline, week 4, and week 8.
  Interventions: Other: Anti-Dynamic Line Cream

INTERVENTIONS:
Other: Anti-Dynamic Line Cream — Topical cream (Formula# 899675 44A) applied to the full face and neck twice daily for 8 weeks. Participants apply 1 g each time in the morning and evening after cleansing, with massage on wrinkle-prone areas. Used after a 2-week wash-out period with standard skincare.

SUMMARY:
The goal of this clinical trial is to find out whether a new cream (Formula# 899675 44A) can help reduce dynamic facial and neck wrinkles in young Chinese women. The main questions it aims to answer are:

* Does the cream lower the appearance of forehead wrinkles, crow's feet, under-eye wrinkles, and nasolabial folds when participants smile or raise their eyebrows?
* Does the cream help reduce horizontal neck folds when participants lower their heads?

About 45 healthy women between the ages of 18 and 35 will take part in this 10-week study. They will:

* Stop using other anti-aging products for 2 weeks (wash-out period)
* Apply the study cream on their face and neck twice a day for 8 weeks
* Visit the clinic 4 times for facial and neck photo collection and clinical assessments
* Learn to make standard facial expressions for photo comparisons

Researchers will compare wrinkle changes using dermatologist scores and photo grading at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese female aged 18-35 years old.
2. All skin types will be contained, including 50% sensitive skin.
3. Regular users of cleanser, anti-aging cream and sunscreen product.
4. Self-claim having concerns of wrinkles problems.
5. Presenting with obvious dynamic wrinkles while making smiling/raising eyebrow expression ( expression reach max condition) evaluated by Dermatologist：

   * Raise eyebrow: Forehead wrinkles (Loreal Atlas, 1<grade≤4)
   * Smile: Underneath eye wrinkles (Loreal Atlas, grade≥3)
   * Smile: Crow's feet wrinkles (Loreal Atlas, grade≥3)
   * Smile: Nasolabial folds (Loreal Atlas, grade>1)
6. Did not participate in any clinical test or cosmetic product test on skin within 3 months.
7. Did not participate any chemical procedures for previous 2 months; and willing to not participate any procedures during the whole study.
8. No disagreement of dermatologist because of other reasons that exclude the participation of the Subject.
9. In general, good health at the time of the study.
10. Willing and able to participate as evidenced by signing of informed consent and photorelease form.
11. Must be willing to comply with all study protocol requirements (pay attention to not take topical or oral treatment like retinol, hormone, antioxidant health-care products which may affect the efficacy of test products).

Exclusion Criteria:

1. Intending to get pregnant, pregnant, lactating or within 6 months of delivery.
2. Subject deprived of rights by a court or administrative order.
3. Major subject to a guardianship order.
4. Subject residing in a health or social care establishment.
5. Patient in an emergency setting.
6. Subject with a skin disease in the test areas (particularly e.g., acne, rosacea, eczema).
7. Subject presenting a stable or progressive serious disease (per investigator's assessment).
8. Immuno-compromised subject.
9. Subject with history of allergy to cosmetic or personal care products or ingredients.
10. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
11. Subjects regularly practicing aquatic or nautical sports.
12. Subjects regularly attending a sauna.
13. Subject with cardiovascular or circulatory history.
14. Subject with a history of skin cancer or malignant melanoma.
15. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Time effect of facial and neck wrinkles (Dermatologist-assessed) | Baseline (T0) to Week 8 (T8wk)
  Clinical scoring of dynamic wrinkles in five facial and neck areas: forehead wrinkles (raising eyebrow), crow's feet wrinkles, underneath eye wrinkles, nasolabial folds (smiling), and horizontal neck folds (lowering head), as assessed by dermatologist at T0, T4wk, and T8wk using the Skin Aging Atlas. Assessment is based on facial expression photos and in-person evaluation. Wilcoxon Signed Rank Test will be used to analyze changes from baseline.

SECONDARY OUTCOMES:
Time effect of facial wrinkles (Expression image-based) | Baseline (T0) to Week 8 (T8wk)
  Dermatologist-assessed wrinkle severity based on a series of 10 expression photos captured at baseline, week 4, and week 8. Areas include forehead wrinkles (raising eyebrow), crow's feet wrinkles, underneath eye wrinkles, nasolabial folds (smiling), and horizontal neck folds (lowering head). Images were taken using DEEP 1.0 and iPhone 15 Pro Max, and graded with the Skin Aging Atlas without referencing prior scores. Statistical analysis used Wilcoxon Signed Rank Test.
Time effect of adverse events and intolerance reactions | Baseline (T0) to Week 8 (T8wk)
  Any reported adverse events (AEs) and local intolerance reactions collected through participant diaries and on-site monitoring at each visit (T0, T4wk, T8wk). All events evaluated for severity, duration, and relation to the test product, and reported within 24 hours per protocol guidelines.
Time effect of product compliance (Twice-daily usage) | Baseline (T0) to Week 8 (T8wk)
  Participant adherence to the instructed regimen of twice-daily application of the investigational cream, assessed by product weight tracking and daily log review at week 4 and week 8 visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon study completion and PRS registration completion.
  Timeline:
  Months 2-3: Data de-identification, metadata preparation, and platform integration.
  Month 4: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn